

# A member of the AstraZeneca Group

# Statistical Analysis Plan

**Protocol Title:** A Phase 1b Study of ACP-196 in Combination with

Obinutuzumab for Patients with Relapsed/Refractory or

Untreated CLL/SLL/PLL

**Protocol Number:** ACE-CL-003

**Sponsor:** Acerta Pharma BV

PPD

5349 AB Oss The Netherlands

**Version / Date:** 

Final: 07 February 2019 Amendment 1: 06 Oct 2021

# A Phase 1b Study of ACP-196 in Combination with Obinutuzumab for Patients with Relapsed/Refractory or Untreated CLL/SLL/PLL

# **Approval Page**

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

| Prepared by: | |
|--------------|-----------------------------|
| PPD | |
| Approval: | |
| PPD | |
| | 07 October 2021 11:58 ADT |
| | Date |
| PPD | |
| | 08 October 2021 15:41 PDT |
| | Date |


# **SAP Revision History:**

| Version/Date | Summary of Major Changes and Rationale |
|---|---|
| Final: 07 February 2019 | New Document |
| Amendment 1: 27 April 2021 | 1. Added Protocol Amendment 7 to Introduction and Overall Study Design sections; updated study schema in accordance with schema updates made in Protocol Amendment 7. |
| | 2. Updated study treatment exposure definitions to cover rituximab and venetoclax. Added definitions for number of cycles administered, dose withholding, and dose reduction. – Section 6.2 |
| | 3. Specified throughout that partial response with lymphocytosis (PRL) is only applicable for Cohorts 1 and 2. |
| | 4. Moved ECOG performance status from Demographics and Baseline Characteristics to Baseline Disease Characteristics. Added "significant fatigue" to the list of B symptoms – Section 10.0 |
| | 5.Added sections 6.1 Prior Anticancer Therapies, 13.2 Adverse Events of Clinical Interest and 13.3 Deaths |
| | 6. Added region and Binet state as demographics and baseline characteristics variables -Section 10.0 |
| | 7.Added infusion interruption and time to the first interruption - Section 6.3 |
| | 8. Moved the ORR at cycle 16 (cohort 3 and 4) from the section of the primary efficacy endpoint to the section of secondary endpoint section -Section 12.1 and 12.2 |
| | 9. Added "nPR(nodular partial remission)" to the definition of DOR(Duration of response) -Section 12.2.4 |
| | 10.Added "time to complete response" and "time to response of PRL or better" – Section 12.2.5 |

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021


# TABLE OF CONTENTS

| TABLE OF CONTENTS | 4 |
|-----------------------------------------------------------------------|----|
| LIST OF ABBREVIATIONS AND DEFINITIONS | 6 |
| 1.0 Introduction | 8 |
| 2.0 Study Objectives | |
| 3.0 OVERALL STUDY design | 9 |
| 4.0 Sample size consideration | 13 |
| 5.0 Analysis POPULATIONS | 15 |
| 5.1 All Treated Population | 15 |
| 5.2 Efficacy Evaluable Population | 15 |
| 6.0 TREATMENTS AND MEDICATIONS | 15 |
| 6.1 Prior Anticancer Therapies | 15 |
| 6.2 Prior and Concomitant Medications | 15 |
| 6.3 Study Treatment Exposure | 16 |
| 7.0 Statistical Methods | 17 |
| 7.1 Data Presentation | 17 |
| 7.2 General Conventions. | 17 |
| 7.3 Analysis Windows | 17 |
| 7.4 Missing Data Handling | 17 |
| 8.0 Subject Disposition | 18 |
| 9.0 Important Protocol deviations | 18 |
| 10.0 demographics and baseline disease characteristics | 18 |
| 11.0 Medical history | 20 |
| 12.0 Efficacy analyses | |
| 12.1 Primary Efficacy Endpoint and Analysis | 20 |
| 12.1.1 Overall Response Rate (ORR) | 20 |
| 12.2 Secondary Efficacy Endpoints and Analyses | |
| 12.2.1 Overall Response Rate(ORR) | |
| 12.2.2 Complete Response Rate and MRD-Negative Complete Response Rate | 21 |
| 12.2.3 Progression-Free Survival | |
| 12.2.4 Duration of Response | 22 |
| 12.2.5 Time to Response | |
| 12.2.6 Time to Next Treatment (TTNT) | 23 |
| 12.2.7 Overall Survival (OS) | 23 |
| 12.2.8 Patient reported outcomes (PRO) | |
| 13.0 Safety Analyses | 25 |
| 13.1 Adverse Events | |
| 13.2 Adverse Events of Clinical Interest. | |
| 13.3 Deaths | |
| 13.4 Laboratory Assessments | 26 |
| 13.4.1 Data Summary Methods | |
| 13.4.2 T/B/NK Cell Counts | 27 |

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

| 13.4.3 Serum Immunoglobulin | 27 |
|---|---|
| 13.4.4 Analysis of Lymphocytosis | |
| 13.5 Vital Signs and Physical Examinations | |
| 13.6 ECOG Performance Status | |
| 14.0 REFERENCE | |
| 15.0 APPENDICES | |
| Appendix A: Analysis Windows | |
| Appendix B: Rai Stage Derivation Criteria | |
| Appendix C: Grading Scale for Hematologic Toxicity in CLL (Hallek 2008) | |
| Appendix D: Defining Prior and Concomitant Medication Flags | 100 |
| Appendix E: Patient Reported Outcomes (PRO) | |
| Appendix F: Adverse Events of Clinical Interest | |

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021


#### LIST OF ABBREVIATIONS AND DEFINITIONS

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021

AE adverse event

AESI adverse event of special interest ALC absolute lymphocyte count ANC absolute neutrophil count

ATC anatomical therapeutic chemical

BID twice per day

BTK Bruton tyrosine kinase CBC complete blood count CI confidence interval

CLL chronic lymphocytic leukemia CR complete remission (response)

CRi CR with incomplete bone marrow recovery

CT computed tomography
DOR Duration of Response
ECI event of clinical interest
ECG electrocardiogram

ECOG Eastern Cooperative Oncology Group

eCRF electronic case report form EDC electronic data capturing

EORTC European Organisation for Research and Treatment of Cancer FACIT-Fatigue Functional Assessment of Chronic Illness Therapy-Fatigue

IGHV immunoglobulin heavy-chain variable

IPD important protocol deviation

IWCLL International Workshop on Chronic Lymphocytic Leukemia

KM Kaplan-Meier

MedDRA Medical Dictionary for Regulatory Activities

mRNA microRNA

MRD Minimal residual disease

NCI-CTCAE National Cancer Institute Common Terminology Criteria for

Adverse Events

nPR nodular partial remission
ORR overall response rate
OS overall survival
PD progression disease
PFS progression-free survival
PLCG2 phospholipase C gamma 2
PLL prolymphocytic leukemia

PK pharmacokinetic

PR partial remission (response)

PRL partial remission (response) with lymphocytosis


| QD | once per day |
|----|--------------|

QD SAE serious adverse event Statistical Analysis Plan SAP

SD stable disease

small lymphocytic lymphoma SLL

sum of the product of the greatest diameters SPD

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

treatment-emergent adverse event **TEAE** 

TNTT time-to-next treatment WHO World Health Organization


#### 1.0 Introduction

This Statistical Analysis Plan (SAP) provides details of the statistical analyses that have been outlined within the protocol for study ACE-CL-003 Protocol Amendment 7 (dated 03 April 2020), which is entitled "A Phase 1b Study of ACP-196 in Combination with Obinutuzumab for Patients with Relapsed/Refractory or Untreated CLL/SLL/PLL."

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021

The original SAP was based on protocol amendment 6 (dated 27 June 2018). The amendment 7 was made to clarify the discontinuation of acalabrutinib might be based on minimal residual disease and clinical response. Also, the protocol was updated to remove the restart of treatment for subjects in treatment-free follow-up to clarify criteria regarding discontinuation and restart of acalabrutinib. The SAP is updated to include changes made in protocol amendment 7.

The scope of the SAP will cover safety and efficacy analyses in ACE-CL-003. Minimal residual disease (MRD), pharmacokinetic (PK), and collection analyses will be provided in the respective reports.

#### 2.0 Study Objectives

The primary objectives are:

#### Cohort 1 and 2:

- To determine the overall response rate (ORR) at 12 months with the combination of acalabrutinib plus obinutuzumab in subjects with relapsed or refractory chronic lymphocytic leukemia (CLL)
- To determine the ORR at 12 months with the combination of acalabrutinib plus obinutuzumab in subjects with treatment-naïve CLL
- To establish the safety and feasibility of the combination of acalabrutinib plus obinutuzumab

#### Cohort 3 and 4:

- To establish the safety of the combination of acalabrutinib plus rituximab plus venetoclax in subjects with relapsed or refractory CLL (Cohort 3)
- To establish the safety of the combination of acalabrutinib plus obinutuzumab plus venetoclax in subjects with treatment-naïve CLL (Cohort 4)

The secondary objectives are:

• To determine the complete response (CR) rate and minimal residual disease (MRD)-negative CR rate in subjects with previously untreated and relapsed and refractory CLL with these regimens (all cohorts)


• To evaluate the ORR of the combination therapy of acalabrutinib plus venetoclax plus an anti-CD20 antibody(rituximab or obinutuzumab) at Cycle 16 (Cohorts 3 and 4)

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

- To determine the time to response, duration of response (DOR), progression-free survival (PFS), time to complete response (CR), time-to-next treatment (TTNT), and overall survival (OS) with these regimens (all cohorts)
- To assess for serial development of resistance by baseline and longitudinal assessment of mutations of Bruton tyrosine kinase (BTK) and phospholipase C gamma 2 (PLCG2) at regular follow-up intervals and by examining diagnosis to relapse samples by whole-exome sequencing (all cohorts)
- To determine trajectory of psychological and behavioral responses to acalabrutinib and covariation with response to therapy (all cohorts)
- To determine the pharmacokinetics of orally administered acalabrutinib (all cohorts) and venetoclax (Cohorts 3 and 4)

The exploratory objectives are:



#### 3.0 OVERALL STUDY design

This is a Phase 1b study with expansion to evaluate the safety and preliminary efficacy of acalabrutinib in combination with obinutuzumab or with venetoclax and an anti-CD20 antibody (rituximab or obinutuzumab) in 4 separate cohorts of subjects: those with relapsed/refractory CLL (Cohorts 1 and 3) and those with treatment-naïve CLL (Cohorts 2 and 4).

A standard 3+3 Phase 1 trial design began in Cohort 1 where the recommended dose was determined. Cohorts 1 and 2 were expanded to better evaluate the toxicity profile of these combination regimens and to detect moderate to large increases in ORR at 12 months relative to historical control. Cohorts 3 and 4 were enrolled to establish the safety profile of the combination of acalabrutinib plus venetoclax plus an anti-CD20 antibody.

For more details on study design, please refer to protocol. Protocol amendments and revision dates are as follows:

Original protocol: 20 May 2014Amendment 1: 28 July 2014


• Amendment 2: 24 March 2015

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

• Amendment 3: 22 July 2015

• Amendment 4: 27 April 2016

• Amendment 5: 03 August 2017

• Amendment 5.1: 06 November 2017

• Amendment 6: 27 June 2018

• Amendment 7: 03 April 2020


#### STUDY SCHEMA

#### PHASE 1B DOSE-ESCALATION PORTION: OBINUTUZUMAB

• At least 6 subjects with relapsed/refractory chronic lymphocytic leukemia (CLL), then at least 6 subjects with treatment-naïve CLL



# **PHASE 1B EXPANSION PORTION**

#### TWO PARALLEL COHORTS ARE TREATED IDENTICALLY

#### COHORT 1:

• Relapsed or refractory disease\*

#### COHORT 2:

- No previous treatment
- 65 years or older OR refuse or are ineligible for approved chemotherapy and/or immunotherapy options



<sup>\*</sup>Samples for pharmacokinetics are obtained from the first 8 subjects enrolled in the Phase 1b expansion of Cohort 1.


<sup>#</sup> Subjects who achieve bone marrow minimal residual disease (MRD)-negative complete response (CR) have the option to discontinue acalabrutinib.

#### STUDY SCHEMA (CONTINUTED)

#### PHASE 1B: COHORTS 3 and 4

Twelve subjects with relapsed/refractory CLL and 12 subjects with treatment-naïve CLL

#### TWO PARALLEL COHORTS ARE TREATED

#### COHORT 3:

• Relapsed or refractory disease\*

#### COHORT 4:

• No previous treatment\*

# ACALABRUTINIB CCI Rituximab CCI Venetoclax CCI



- \*Samples for pharmacokinetics are obtained from the first 8 subjects enrolled in each of Cohorts 3 and 4.
- <sup>#</sup> Discontinuation of acalabrutinib after collection is possible by investigator decision based on minimal residual disease (MRD) and clinical response (refer to the Schedule of Assessments in Table 12 and 13 of the protocol).


#### 4.0 Sample size consideration

The sample size for Cohorts 1 and 2 is based on: 1) dose de-escalation rules and 2) the number of subjects required to detect moderate to large increases in ORR relative to historical control with sufficient power while constraining Type I error to 0.10. This study is expected to require 45 subjects, 6 subjects evaluated for safety in each cohort and an additional 20 and 13 subjects enrolled in Cohorts 1 and 2, respectively. More subjects may be enrolled if de-escalation of dose levels is indicated in the safety evaluation.

Protocol: ACE-CL-003 Amendment 1: 27 April 2021

The sample size of 12 subjects each for Cohorts 3 and 4 is chosen to provide evaluation for safety and tolerability.

#### Cohorts 1 and 2

Each of Cohorts 1 and 2 are expanded at the recommended dose level to include, respectively, 26 and 19 total relapsed/refractory and treatment-naïve CLL subjects. These sample sizes were chosen to obtain sufficient preliminary safety and efficacy information in these populations. With respect to toxicity and ability to detect common adverse events (AEs), there is an approximately 60% chance of observing at least 1 subject with an AE occurring at a 5% rate with 19 treatment-naïve subjects in Cohort 2 and an approximately 75% chance in the group of 26 relapsed/refractory CLL subjects in Cohort 1.

If toxicity profiles are similar and it is appropriate to summarize AEs across all subjects, there is at least a 90% chance of detecting a common AE. With respect to clinical efficacy, a 50% ORR (partial response with lymphocytosis or better) (null) at the 12-month evaluation would be considered uninteresting because this can be achieved with either acalabrutinib or obinutuzumab as single agents in both populations. However, an ORR of at least 75% in the relapsed/refractory setting for Cohort 2 and an ORR of at least 80% in the treatment-naïve setting for Cohort 1 would be of considerable interest and would warrant further investigation of the combination regimen (alternative).

If 16 or fewer responses are observed in 26 evaluable subjects with relapsed/refractory CLL in Cohort 1, the combination of acalabrutinib with obinutuzumab would not be considered promising; likewise, if 12 or fewer responses in 19 evaluable subjects who were previously untreated for CLL in Cohort 2 were observed, the combination would not be considered promising as upfront therapy. Each of these designs has at least 90% power with a one-sided alpha level of 0.10.

#### Cohorts 3 and 4

The sample sizes for Cohorts 3 and 4 are chosen to obtain preliminary safety information in the relapsed/refractory and treatment-naïve CLL populations. With respect to toxicity and ability to detect common AEs, there is a 46% chance of observing at least 1 subject with an AE occurring at a 5% rate with 12 subjects in each of Cohorts 3 and 4.


Below is a list of various AE rates with the chance of observing in at least 1 subject.

| Sample Size | Adverse Event Rate | Chance of Observing at Least 1 Adverse Event |
|---|---|---|
| 12 | 1% | 11% |
| 12 | 2% | 22% |
| 12 | 5% | 46% |
| 12 | 10% | 72% |

Protocol: ACE-CL-003

Amendment 1: 27 April 2021


#### **5.0 Analysis POPULATIONS**

Analysis populations will be defined in the following sections. The efficacy and safety analyses will be performed on the All Treated Population. The primary efficacy analysis will be based on the Efficacy Evaluable Population.

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

#### 5.1 All Treated Population

The All Treated Population will include all enrolled subjects who received ≥1 dose of study drug.

All enrolled subjects were treated with at least one dose of study drug in this study, thus all-treated population is the same as the enrolled population.

#### 5.2 Efficacy Evaluable Population

The Efficacy Evaluable Population will include all subjects in the All Treated Population who had ≥1 response assessment after the first dose of study drug.

#### 6.0 TREATMENTS AND MEDICATIONS

#### **6.1 Prior Anticancer Therapies**

A prior anticancer therapy is defined as a systemic therapy subjects received, either as a single or combination therapy, for the treatment of active CLL/SLL with an end date occurring before the date of first dose of study treatment. Therapies given as a consolidation or maintenance of a response or remission will not be considered as a separate regimen. The number of prior therapies, type of prior therapy, and time (months) from the end of last therapy to the first dose of study drug will be summarized.

#### **6.2 Prior and Concomitant Medications**

Prior and concomitant medications will be coded according to the World Health Organization (WHO) drug dictionary. Medications started or ended prior to first dose will be considered as prior medications. Concomitant medication is defined as all medications used on or after the first dose, through the treatment phase, and for 30 days following the last dose of study drug. With use of this definition, a medication can be classified as both prior and concomitant. Medications with completely missing start and stop dates will be considered as both prior and concomitant medications.

Appendix D shows the prior and concomitant medication flags for various scenarios. The number and percentage of subjects will be presented by anatomical therapeutic chemical (ATC) classification system Level 2 and preferred term.


Prior and concomitant medications will be summarized by the WHO drug dictionary Anatomical Therapeutic Chemical (ATC) level 2 and preferred term (PT).

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

## **6.3 Study Treatment Exposure**

Study treatment exposure will be summarized for all subjects in the Safety population. The following will be provided for each treatment component when applicable:

- Duration of exposure
  - Acalabrutinib and venetoclax (months): (last dose date first dose date + 1) / 30.4375
  - Obinutuzumab and rituximab (days): (last dose date first dose date + 28)
- Cumulative dose received on study (acalabrutinib, venetoclax, rituximab, and obinutuzumab)
- Average daily dose (acalabrutinib and venetoclax only)
  - Calculated as (total dose received [mg] / duration of exposure [days])
- Relative dose intensity
  - Acalabrutinib:
  - Calculated as (total cumulative dose received [mg] / (duration of exposure [days] \*
  - 100 [mg] \* 2) \*100)
  - Obinutuzumab:
  - Calculated as (total volume infused (mg) / 8000 mg \* 100)
  - Rituximab:
  - Calculated as (total dose infused [mg] / total cumulative planned dose based on
  - body surface area  $[375 \text{ mg/m}^2] * 100$
  - Venetoclax:
  - Calculated as (total cumulative dose received [mg] / 136,990 mg \* 100)
- Dose withholding
  - Acalabrutinib: missing dose for  $\geq 7$  consecutive days
  - Venetoclax, Obinutuzumab, Rituximab: missing dose for at least 1 day
- Dose reduction
  - Acalabrutinib: taking lower dose level for  $\geq 3$  consecutive days
  - Venetoclax, Obinutuzumab, Rituximab: taking lower dose level for at least 1 day
- Infusion interruption (Obinutuzumab and Rituximab only)


• Time to first interruption (days) (Obinutuzumab and Rituximab only)

#### 7.0 Statistical Methods

#### 7.1 Data Presentation

Tables and figures will be summarized by cohort unless otherwise specified.

No formal tests of hypotheses will be performed. P-values, if presented, will be provided for descriptive purpose. Descriptive statistics (number of subjects, mean, and standard deviation, median, minimum, and maximum) will be presented for continuous variables, including baseline demographic, disease characteristics, study drug administration, efficacy and safety outcomes. Categorical variables will be summarized as the number and percentage of subjects per category. Confidence intervals [CIs] may be included as appropriate.

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

#### 7.2 General Conventions

<u>Baseline</u> is defined as the last measurement taken prior to the first dose of study drug administration. <u>Post-baseline</u> is defined as a measurement taken after the first dose of study drug administration.

<u>Study Day 1</u> is defined as the date of first dose. For visits (or events) that occur on or after first dose date, study day is calculated as (date of visit [event] – date of first dose + 1). For visits (or events) that occur prior to first dose date, study day is calculated as (date of visit [event] – date of first dose). There is no Study Day 0.

Laboratory data summary will be based on central laboratory results. Local laboratory results will be used if central laboratory results are not available. Central laboratory results will use reference ranges provided by the central laboratory, and local laboratory results will use the reference ranges provided by local laboratories.

#### 7.3 Analysis Windows

For parameters summarized by visit, an analysis window will be assigned to each nominal visit. Each assessment will be assigned to an analysis visit based on the analysis window in which the assessment date falls. Details are defined in Appendix A.

#### 7.4 Missing Data Handling

No imputation for missing values of efficacy endpoints. Imputation for missing dates such as AE start or end dates and prior and concomitant medication start dates or end dates will be documented in the programming specifications.


#### 8.0 Subject Disposition

Subject disposition will present the number and percentage of subjects in All Treated Population and Efficacy Evaluable Population, who discontinue treatment and reasons, and who do not complete the Safety follow-up as well as the reasons, time on treatment, and time on study.

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021

#### 9.0 Important Protocol deviations

Important protocol deviation (IPD) categories are defined and managed by the study team during the IPD reviews throughout the study before database lock. These definitions of IPD categories, subcategory codes, and descriptions will be used during the course of the study. The final IPD list is used to produce the summary table and by-subject listing for IPDs.

#### 10.0 demographics and baseline disease characteristics

The following variables collected at baseline will be presented:

- Demographics and baseline characteristics
  - Age (years)
    - Descriptive statistics
    - o <65 vs. ≥65 years
    - $\circ$  <70 vs.  $\geq$ 70 years
  - Sex (male, female)
  - Race
    - o American Indian/Alaskan Native, African American/Black, Asian, Caucasian/White, Native Hawaiian/Other Pacific Islander or Other
  - Ethnicity (Hispanic or Latino, Non-Hispanic or Latino)
  - Height
  - Weight
  - Region (single site, United States)
  - ECOG performance status
- ➤ Baseline disease characteristics
  - Histology
    - o For RR, TN
      - CLL
      - SLL


- PLL
- Time since initial CLL diagnosis to first dose (years)
- Rai stage Rai stage collected on the electronic case report form (eCRF) and derived Rai stage based on variables collected at screening visit using the criteria described in Appendix B

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

- Bulky disease (not applicable for RS/PLL) defined as if at least one dimension of the lymph node measurement is
  - o ≥5 cm
  - o ≥10 cm
- B symptoms weight loss, fever, night sweats, significant fatigue
- Chromosomal abnormalities
  - o del(17)(p13.1) (TP53)
  - o del(11)(q22.3) (ATM)
- β2-microglobulin
  - $\circ$  >3.5 vs.  $\leq$ 3.5 mg/L
  - $\circ$  >3 vs.  $\leq$ 3 mg/L
- Number of prior systemic therapy
  - Descriptive statistics
  - $\circ$  <3 vs.  $\geq$ 3
- Type of prior systemic therapy
- Time since most recent therapy (months)
- Cytopenia
  - Absolute neutrophil count (ANC)  $\leq 1.5 \times 10^{9}$ /L
  - o Hemoglobin ≤11g/dL
  - $\circ$  Platelet  $\leq 100 \times 10^{9} / L$
  - Hemoglobin  $\leq 11$ g/dL or platelet  $\leq 100$ x10 $^9$ /L
  - o Any of the above
- ANC (10^9/L)
- Absolute lymphocyte count (ALC) (10^9/L)
- Hemoglobin (g/dL)


- Platelets (10^9/L)
- IGHV mutation status (Unmutated IgHV, Mutated IgHV)
- ZAP-70 Methylation Status (Positive, Negative, Not Done/NA)

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

- Complex Karyotype
  - o Subjects with complex karyotype
  - o Subjects without complex karyotype

#### 11.0 Medical history

Medical history data will be coded per the Medical Dictionary for Regulatory Activities (MedDRA), summarized by system organ class and preferred term, and presented as a data listing

#### 12.0 Efficacy analyses

Response will be assessed by investigators based on International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Response Assessment Criteria (modified from Hallek 2008) with incorporation of the clarification for treatment-related lymphocytosis per Cheson 2012 for CLL/SLL.

The efficacy analysis will be performed using All Treated Population. The Efficacy Evaluable Population will be used for primary efficacy analysis.

#### 12.1 Primary Efficacy Endpoint and Analysis

#### 12.1.1 Overall Response Rate (ORR)

ORR is the proportion of subjects who achieve complete remission (CR), CR with incomplete bone marrow recovery (CRi), nodular partial remission(nPR), or partial remission (PR) while on treatment before the initiation of new anticancer therapy or stem cell transplant.

For Cohorts 1 and 2, the ORR(PR or better) at the all available response assessments up to the 12-months will be calculated and 95% exact binomial CIs will be provided.

ORR will be summarized using All Treated Population and Efficacy Evaluable Population.

For CLL disease subgroups, ORR, including PRL as a response, (only for Cohorts 1 and 2), will also be summarized in the same fashion.

#### 12.2 Secondary Efficacy Endpoints and Analyses

The secondary efficacy analyses will be performed using All Treated Population.


### 12.2.1 Overall Response Rate(ORR)

The ORR of the combination therapy of acalabrutinib plus venetoclax plus an anti-CD20 antibody at Cycle 16 (Cohorts 3 and 4) will be calculated and 95% exact binomial CIs will be provided

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021

#### 12.2.2 Complete Response Rate and MRD-Negative Complete Response Rate

The CR rate will be calculated and corresponding 95% confidence intervals through use of exact binomial distribution will be provided. The MRD-Negative CR rate will be summarized with MRD data in separate report..

# 12.2.3 Progression-Free Survival

PFS is defined as the time from the date of first dose to the date of first disease progression or death due to any cause, whichever comes first. If no disease progression or death is reported for a subject, the subject will be censored at the date of last adequate assessment (censoring date). If a subject receives an autologous or allogeneic stem cell transplant, the subject will be censored at the date of transplant. If a subject starts new anticancer therapy before disease progression or death, the subject will be censored at the date of last adequate assessment prior to receiving the new anticancer therapy. Adequate assessment is defined as physical examination (PE) and complete blood count (CBC) or computed tomography (CT) for CLL disease subgroups (or PET-CT for RS/PLL disease subgroup) and CBC. If a subject does not have any adequate assessment after first dose, the subject will be censored at Day 1.

PFS is calculated as date of disease progression or death (or censoring date for censored subjects) - first dose date + 1.

Events and censoring rules for PFS are summarized as follows:

| Situation | Outcome | Date | Event Description/<br>Censoring Reason |
|---|---|---|---|
| Documented Progression of Disease (PD) | Event | Earliest date of<br>disease<br>assessment<br>documenting PD | PD |
| Death | Event | Date of Death | Death |
| Start of new anticancer therapy before documented PD or death | Censored | Date of last<br>adequate<br>assessment prior<br>to receiving the<br>new anticancer<br>therapy | New anticancer<br>therapy |


| Start of transplant | Censored | Date of transplant | Transplant |
|---|---|---|---|
| Withdrawal of consent before documented PD or death | Censored | Date of last<br>adequate disease<br>assessment | Withdrawal of consent |
| Lost to follow-up before documented PD or death | Censored | Date of last<br>adequate disease<br>assessment | Lost to follow-up |
| No documented PD or death and the reason for not completing Safety Follow-up visit is "Other" | Censored | Date of last<br>adequate disease<br>assessment | Other: specify |
| No documented PD or death at the time of data cutoff | Censored | Date of last<br>adequate disease<br>assessment | Data cutoff |
| No post-baseline adequate disease assessments | Censored | Date of first dose | No post-baseline<br>adequate disease<br>assessments |

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021

Kaplan-Meier (KM) curve will be used to estimate the distribution of PFS. Median PFS and the 95% confidence limits and PFS rates for selected landmarks with 95% CIs will be reported. Number of progressions, deaths, and censored events by reason will be summarized.

#### 12.2.4 Duration of Response

Duration of response (DOR) is defined as the time from the date of achieving the first CR, CRi, nPR, or PR to the date of disease progression or death due to any cause, whichever comes first. Subjects who do not experience a disease progression or death will be censored using the same rule for PFS as described in Section 12.2.3.

DOR is calculated as date of disease progression or death (or censoring date for censored subjects) – date of achieving the first CR, CRi, nPR or PR + 1.

DOR will be analyzed similarly to PFS including a KM plot, as described in section 12.2.3.

#### 12.2.5 Time to Response

The following time to response will be calculated and summarized using descriptive statistics.

- Time to CR = (date of CR date of first dose +1)/30.4376
- Time to CR/CRi = (date of first CR or CRi date of first dose +1)/30.4376
- Time to response of PR or better = (date of first PR or better date of first dose + 1) / 30.4376


-

• Time to response of PRL or better = (date of first PRL or better – date of first dose + 1) / 30.4376

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

#### 12.2.6 Time to Next Treatment (TTNT)

TTNT is defined as the time from the date of first dose to the date of institution of subsequent anticancer therapy for CLL or death due to any cause, whichever comes first. Subjects who do not have the above-specified events prior to the data cutoff date will be censored at the date of last visit. TTNT will be calculated as: (Earlier date of institution of subsequent anticancer therapy for CLL or death due to any cause) – date of first treatment + 1. For censored subjects, date of last visit will replace earlier date of use of subsequent anticancer therapy for CLL or death due to any cause in the calculation.

TTNT will be analyzed similarly to PFS including a KM plot, as described in section 12.2.3.

#### 12.2.7 Overall Survival (OS)

Overall survival (OS) is defined as the time from the date of first doseto death due to any cause. Subjects who were not known to have died prior to the analysis data cutoff date will be censored as follows:

| Situation | Outcome | Date | Event Description/<br>Censoring Reason |
|---|---|---|---|
| Death on or before data cutoff | Event | Date of death | Death |
| Exit study prior to data cutoff | Censored | Date of<br>discontinuation<br>from study<br>participation as<br>reported on study<br>exit CRF | Withdrew consent/<br>study terminated by<br>sponsor/study exit |
| Lost to follow-up prior to data cutoff | Censored | Date subject last known to be alive | Lost to follow-up |
| No death reported on or before data cutoff | Censored | Date subject last known to be alive | Still on study |

OS will be calculated as death date (or censoring date) – the date of first dose + 1.

OS will be analyzed similarly to PFS including a KM plot, as described in section 12.2.3.

#### 12.2.8 Patient reported outcomes (PRO)

The patient reported outcomes include:

• The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) is a 30-item questionnaire designed to assess health-


related quality of life in cancer patients. There are 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 3 symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale. Several single-item symptom measures are also included (dyspnea, insomnia, appetite, constipation, diarrhea, and financial impact).

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021

• Medical outcomes Study Short Form 36 (SF-36) is used to assess health-related quality of life. It consists of eight scales (physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health) yielding two summary measures: physical and mental health

EORTC QLQ-C30 and SF36 will be collected at screening, Cycle 5, Cycle 9, Cycle 13, Cycle 18, Cycle 24 and end of study.

#### Cohorts 1 and 2:

Cohorts 1 and 2 collected EORTC QLQ-C30 and SF-36 and they are used to assess patient-reported quality of life.

Mean in mental/physical component scale for SF36, and each item of symptoms/functioning /global health status for EORTC QLQ-C30 is calculated at baseline and cycle 24. A repeated measures ANOVA is used to assess quality of life across the study period, using baseline and 24-month outcomes. Cohort (treatment-naïve and relapsed/refractory) is the factor used among patients to assess time-related outcomes and to determine any cohort, time, and interaction effects for individual patients.

The analyses were performed by Ohio State University Comprehensive Cancer Center and the results were published in the journal Cancer Discovery [5].

#### Cohorts 3 and 4:

Cohorts 3 and 4 collected EORTC QLQ-C30 only and is used to measure quality of life in cancer patients. The Sponsor will perform analysis to summarize EORTC QLQ-C30 for Cohorts 3 and 4.

The EORTC QLQ-C30 scale scores will be calculated using the EORTC QLQ-C30 Scoring Manual (Fayers & et al, 2001). The instrument yields the following scales:

- Global health status / Quality of Life (QoL) (2 items)
- Functional scales
  - Physical functioning (5 items)


- o Role functioning (2 items)
- o Emotional functioning (4 items)
- o Cognitive functioning (2 items)
- o Social functioning (2 items)
- Symptom scales / items
  - o Fatigue (3 items)
  - o Nausea and vomiting (2 items)
  - o Pain (2 items)
  - Dyspnea, insomnia, appetite loss, constipation, diarrhea, Financial impact (1 item each)

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021

The principle for scoring is the same for all scales. In brief, outcome scores are computed by standardizing the average of the items (i.e., a raw score) making up the scale. Outcome scores are computed using a linear transformation of the raw score such that scores range from 0 to 100. Details are provided in Appendix E: Patient Reported Outcomes (PRO). A higher score represents a higher ("better") level of functioning or a higher ("worse") level of symptoms; that is, a high score for a functional scale represents a high/healthy level of functioning, a high score for the GHS represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems. Note that the global health status scale is based on only the 2 specific HRQoL items and not the entire questionnaire.

If at least half the items of a scale are present for a time point, then the score will be calculated using the average of all items answered; otherwise, the score will be set to missing. For single measures, if the item is missing the scale score is set to missing.

Baseline is defined as the last available record on or prior to the start date of study treatment.

At each analysis visit and for cohort, the summary statistics (number of subjects, mean, standard deviation, median, and range) of scaled scores and changes from baseline scale scores will be calculated for global health status/QoL, each functional scale and each symptom scale by cohort at each analysis visit.

A listing of scale scores will be generated. A mean overtime plot will be generated for the global health status/quality of life. Also, the compliance to the schedule of administration will be summarized by cohort for baseline and post-baseline timepoints.

#### 13.0 Safety Analyses

Safety analyses will be performed using the All Treated Population unless specified otherwise.

Safety will be assessed by evaluation of treatment-emergent adverse events (TEAEs), laboratory values, vital signs measurements, electrocardiogram (ECG) results, physical examinations, and Eastern Cooperative Oncology Group (ECOG) performance status.


#### 13.1 Adverse Events

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA v 24.0) reporting system. The investigator will grade AEs according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03 for AEs. Hematologic toxicity is assessed by the investigator according to IWCLL 2008 guidelinesfor Cohorts 1 and 2, and NCI CTCAE v4.03 for Cohorts 3 and 4. TEAEs are defined as those events that occur on or after the first dose of study drug, through the treatment phase, and within 30 days following the last dose of study drug.

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021

All TEAEs will be summarized by cohort as treated. For each cohort, AE incidence rates will be summarized with frequency and percentage by system organ class and preferred term, and the denominator for the AE incidence rate will be based on the number of subjects treated in that cohort unless otherwise specified. In addition, AE incidence rates will also be summarized by severity. and relationship to study drug. Relationship to study drug, per the investigator's judgment, is recorded on the CRF.

Subjects with multiple occurrences of events for a given preferred term, system organ class, or overall will be counted only once at the maximum severity. and strongest relationship to study drug for each preferred term, system organ class, and overall, respectively.

Summaries will be presented for:

- treatment-emergent AEs
- treatment-emergent serious adverse events (TESAEs)
- treatment-related TEAEs
- treatment-related TESAEs
- AEs leading to study drug discontinuation or dose modifications or dose delay
- treatment-emergent fatal (Grade 5) AEs

#### 13.2 Adverse Events of Clinical Interest.

Adverse events of clinical interest(ECIs) are specified in Appendix F. Subject incidence rates of AEs of clinical interest will be summarized similarly to TEAEs by cohort.

#### 13.3 Deaths

All reported deaths will be summarized by cohort and cause of death. A by-subject listing that includes date of death and cause of death will be provided.

#### 13.4 Laboratory Assessments

#### 13.4.1 Data Summary Methods

All laboratory values will be converted to and reported as SI units and classified as normal, low, or high based on the normal ranges provided by the local laboratory.


Hematologic parameters, including platelet counts, hemoglobin, and neutrophils, will be summarized by IWCLL 2008 (Appendix C) and NCI CTCAE v4.03 respectively. All other gradable laboratory parameters will be graded using the NCI CTCAE v4.03.

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

Per the grading scale in the IWCLL guidelines, ANC: Both baseline grade and post-baseline grade are defined based on absolute values and 2) Hemoglobin and platelet: baseline grade is not applicable (no criterion is provided to define baseline grade) and post-baseline grade is based on percentage decrease from baseline value.

Gradable parameters that have criteria available for both low and high values (e.g., hypercalcaemia for a high value of calcium and hypocalcaemia for a low value of calcium) based on the NCI CTCAE v4.03 will be summarized for both criteria (low and high). Subjects will be counted only once for each criterion/direction. The same subject can be counted for both criteria if the subject has laboratory values meeting each criterion. Subjects meeting the criteria for Grade 1 or higher for the high direction will be summarized under Grade 0 when summarizing the low direction and vice versus.

For each laboratory parameter, the baseline laboratory value/grade is defined as the last laboratory value/grade collected on or prior to the date of the first dose of study drug. The change from baseline to post-baseline value will be calculated for each parameter.

#### 13.4.2 T/B/NK Cell Counts

Descriptive statistics will be presented at baseline, last post-baseline, minimum post-baseline, and maximum post-baselinefor the flow cytometry testing parameters (CD3<sup>+</sup>, CD4<sup>+</sup>, CD8<sup>+</sup>, CD19<sup>+</sup>, and NK cells).

Changes from baseline at each of the last, minimum, and maximum post-baseline time points will be summarized. Figures will be presented for the mean of selected parameters over time as appropriate.

#### 13.4.3 Serum Immunoglobulin

For IgG, IgM, and IgA levels, descriptive statistics will be presented at baseline, last post-baseline, minimum post-baseline, and maximum post-baseline. Changes from baseline at each of the last, minimum, and maximum post-baseline time points will be summarized. Figures will be presented for the mean of selected parameters over time as appropriate.

#### 13.4.4 Analysis of Lymphocytosis

Lymphocytosis is defined as an elevation in ALC of  $\geq 50\%$  compared with baseline and a post-baseline assessment  $\geq 5,000/\mu L$ .

The number, percentage (and 95% exact binomial CI) of subjects with at least once occurrence of lymphocytosis will be summarized.


Time to Lymphocytosis will be calculated from the date of the first dose of study drug to the first post-baseline ALC which met the lymphocytosis criteria and summarized using descriptive statistics.

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

Duration of lymphocytosis (DOL) is defined as the duration of time from the earliest date on which the ALC value met the lymphocytosis criteria at a post-baseline assessment to the earliest date on which a subsequent ALC value met the resolution criteria. Resolution of lymphocytosis is defined as 1) a decrease of ALC value to the baseline level or lower or 2) an achievement of ALC value that is below  $5,000/\mu$ L, whichever occurs first.

DOL = Earliest date of meeting resolution criteria - Earliest date of meeting lymphocytosis criteria + 1.

Confirmation is not required for resolution of lymphocytosis. Subjects who developed lymphocytosis but whose lymphocytosis was not resolved prior to the analysis cutoff date will be censored at the last sample date with non-missing ALC value at or prior to the analysis cutoff date. KM curves will be used to estimate the distribution of DOL. The 50th percentile of KM estimates along with its two-sided 95% CI will be used to estimate the median DOL.

#### 13.5 Vital Signs and Physical Examinations

For each vital sign measurement, descriptive statistics will be presented at baseline, last post-baseline, minimum post-baseline, and maximum post-baseline. Change from baseline at each of the last, minimum, and maximum post-baseline time points will be summarized.

Findings of abnormal physical examinations at baseline and post-baselinewill be tabulated by body system at each visit.

Shift of blood pressure from baseline to the worst score during the treatment will be provided as shift tables.

#### 13.6 ECOG Performance Status

Shift of ECOG from baseline to the worst score during the treatment will be summarized in a shift table.

#### 14.0 REFERENCE

- [1] Byrd JC, Furman RR, Coutre SE, et al. Targeting Btk with ibrutinib in relapsed chronic lymphocytic leukemia. N Engl J Med 2013;369:32-42. Erratum in: N Engl J Med 2014b;370:786.
- [2] Cheson BD, Byrd JC, Rai KR, et al. R novel targeted agents and the need to refine clinical end points in chronic lymphocytic leukemia. J Clin Oncol 2012;30:2820-2.


[3] Cheson BD, Fisher RI, Barrington SF, et al. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: The Lugano Classification. J Clin Oncol 2014;32:3059-68.

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

- [4] Hallek M, Cheson BD, Catovsky D, et al. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood 2008;111:5446-56.
- [5] Jennifer A. Woyach, James S. Blachly, Kerry A. Rogers, et al. Acalabrutinib plus Obinutuzumab in Treatment-Naïve and Relapsed/Refractory Chronic Lymphocytic Leukemia. *Cancer Discovery* 2020;10:394-405.

#### 15.0 APPENDICES

**Appendix A: Analysis Windows** 

| Tumor assessment/CT/SPD For Cohort 1 and 2 | | | | |
|---|---|---|---|---|
| | | | Analysis Window<br>(Study Day) | |
| Nominal<br>Visit | Study<br>Day | Nominal<br>Month | Lower<br>(inclusive) | Upper (inclusive) |
| C4D1 | 85 | 0 | | 127 |
| C7D1 | 169 | 1 | 128 | 211 |
| C10D1 | 253 | 1 | 212 | 281 |
| C12D1 | 309 | 1 | 282 | 351 |
| C15D1 | 393 | 13 | 352 | 435 |
| C18D1 | 477 | 15 | 436 | 519 |
| C21D1 | 561 | 18 | 520 | 603 |
| C24D1 | 645 | 21 | 604 | 687 |
| C30D1 | 813 | 27 | 688 | 855 |
| C36D1 | 981 | 32 | 856 | |


| Tumor assessment/CT/SPD For Cohort 3 and 4 | | | | |
|---|---|---|---|---|
| | | | Analysis Window<br>(Study Day) | |
| Nominal<br>Visit | Study<br>Day | Nominal<br>Month | Lower (inclusive) | Upper (inclusive) |
| C4D1 | 85 | 0 | | 127 |
| C7D1 | 169 | 1 | 128 | 211 |
| C10D1 | 253 | 1 | 212 | 295 |
| C13D1 | 337 | 1 | 296 | 379 |
| C16D1 | 421 | 13 | 380 | 463 |
| C19D1 | 505 | 15 | 464 | 547 |
| C22D1 | 589 | 18 | 548 | 617 |
| C24D1 | 645 | 21 | 618 | 687 |
| C30D1 | 813 | 27 | 688 | 855 |
| C36D1 | 981 | 32 | 856 | |

| Hematology / Chemistry | | | | |
|---|---|---|---|---|
| | | | Analysis Window<br>(Study Day) | |
| Nominal<br>Visit | Study<br>Day | Nominal<br>Month | Lower (inclusive) | Upper (inclusive) |
| C1D1 | 1 | 0 | | 1 |
| C1D8 | 8 | 1 | 2 | 12 |
| C1D15 | 15 | 1 | 13 | 21 |
| C2D1 | 29 | 1 | 22 | 43 |
| C3D1 | 57 | 2 | 44 | 71 |
| C4D1 | 85 | 2 | 72 | 99 |
| C5D1 | 113 | 3 | 100 | 127 |
| C6D1 | 141 | 4 | 128 | 155 |
| C7D1 | 169 | 5 | 156 | 183 |
| C8D1 | 197 | 6 | 184 | 211 |
| C9D1 | 225 | 7 | 212 | 239 |
| C10D1 | 253 | 8 | 240 | 267 |
| C11D1 | 281 | 9 | 268 | 295 |
| C12D1 | 309 | 10 | 296 | 351 |
| C15D1 | 393 | 13 | 352 | 435 |


Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

| C18D1 | 477 | 15 | 436 | 519 |
|-------|-----|----|-----|-----|
| C21D1 | 561 | 18 | 520 | 603 |
| C24D1 | 645 | 21 | 604 | 687 |
| C30D1 | 813 | 27 | 688 | 855 |
| C36D1 | 981 | 32 | 856 | |

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

| Physical Examination/ECOG | | | | |
|---|---|---|---|---|
| | | | Analysis (Study | |
| Nominal<br>Visit | Study<br>Day | Nominal<br>Month | Lower (inclusive) | Upper (inclusive) |
| C1D1 | 1 | 0 | | 1 |
| C1D8 | 8 | 1 | 2 | 12 |
| C1D15 | 15 | 1 | 13 | 21 |
| C2D1 | 29 | 1 | 22 | 43 |
| C3D1 | 57 | 2 | 44 | 71 |
| C4D1 | 85 | 2 | 72 | 99 |
| C5D1 | 113 | 3 | 100 | 127 |
| C6D1 | 141 | 4 | 128 | 155 |
| C7D1 | 169 | 5 | 156 | 183 |
| C8D1 | 197 | 6 | 184 | 211 |
| C9D1 | 225 | 7 | 212 | 239 |
| C10D1 | 253 | 8 | 240 | 267 |
| C11D1 | 281 | 9 | 268 | 295 |
| C12D1 | 309 | 10 | 296 | 351 |
| C15D1 | 393 | 13 | 352 | 435 |
| C18D1 | 477 | 15 | 436 | 519 |
| C21D1 | 561 | 18 | 520 | 603 |
| C24D1 | 645 | 21 | 604 | 687 |
| C30D1 | 813 | 27 | 688 | 855 |
| C36D1 | 981 | 32 | 856 | |


| Stage | Lymphocytosis | Lymphadenopathy | Hepatomegaly or splenomegaly | Anemia | Thrombocytopenia |
|---|---|---|---|---|---|
| 0 | 1 | 0 | 0 | 0 | 0 |
| Ι | 1 | 1 | 0 | 0 | 0 |
| II | 1 | any | 1 | 0 | 0 |
| III | 1 | any | any | 1 | 0 |
| IV | 1 | any | any | any | 1 |

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021


<sup>1 =</sup> yes, 0 = no, any = yes or no

#### **Appendix C: Grading Scale for Hematologic Toxicity in CLL (Hallek 2008)**

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

| | Decrease in platelets <sup>2</sup> or | A1 1t |
|---|---|---|
| | Hb <sup>3</sup> (nadir) from | Absolute neutrophil |
| Grade <sup>1</sup> | pretreatment value | count/μL <sup>4</sup> (nadir) |
| 0 | No change to 10% | ≥2000 |
| 1 | 11%-24% | ≥1500 and <2000 |
| 2 | 25%-49% | $\geq$ 1000 and $<$ 1500 |
| 3 | 50%-74% | ≥500 and <1000 |
| 4 | ≥75% | < 500 |

- 1. Grades: 1, mild; 2, moderate; 3, severe; 4, life-threatening; 5, fatal. Death occurring as a result of toxicity at any level of decrease from pretreatment will be reported as Grade 5.
- 2. Platelet counts must be below normal levels for Grades 1 to 4. If, at any level of decrease, the platelet count is <20 x 10<sup>9</sup>/L (20,000/μL), this will be considered Grade 4 toxicity, unless a severe or life-threatening decrease in the initial platelet count (e.g., <20 x 10<sup>9</sup>/L [20,000/μL]) was present pretreatment, in which case the patient is not evaluable for toxicity referable to platelet counts.
- 3. Hemoglobin (Hb) levels must be below normal levels for Grades 1 to 4. Baseline and subsequent Hb determinations must be performed before any given transfusions. The use of erythropoietin is irrelevant for the grading of toxicity but should be documented.
- 4. If the ANC reaches <1 x 10<sup>9</sup>/L (1000/μL), it should be judged to be Grade 3 toxicity. Other decreases in the white blood cell count or in circulating neutrophils are not to be considered because a decrease in the white blood cell count is a desired therapeutic endpoint. A gradual decrease in granulocytes is not a reliable index in CLL for stepwise grading of toxicity. If the ANC was <1 x 10<sup>9</sup>/L (1000/μL) before therapy, the patient is not evaluable for toxicity referable to the ANC. The use of growth factors such as granulocyte colony-stimulating factor (G-CSF) is not relevant to the grading of toxicity but should be documented.


# **Appendix D: Defining Prior and Concomitant Medication Flags**

The figure below depicts various scenarios of prior and concomitant medications. The prior and concomitant medication flags are specified respectively for each scenario.

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021



- 1 = start < first dose and stop < first doe
- = start < first dose and stop >= first dose
- 3 =start >= first dose
- 4 = start > last dose + 30 days


# **Appendix E: Patient Reported Outcomes (PRO)**

## 1. EORTC QLQ-C30

The United States English version is provided as an example only.



# EORTC QLQ-C30 (version 3)

We are interested in some things about you and your health. Please answer all of the questions yourself by circling the number that best applies to you. There are no "right" or "wrong" answers. The information that you provide will remain strictly confidential.

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

Please fill in your initials:
Your birthdate (Day, Month, Year):
Today's date (Day, Month, Year):
31

| | | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|---|
| 1. | Do you have any trouble doing strenuous activities,<br>like carrying a heavy shopping bag or a suitcase? | 1 | 2 | 3 | 4 |
| 2. | Do you have any trouble taking a <u>long</u> walk? | 1 | 2 | 3 | 4 |
| 3. | Do you have any trouble taking a short walk outside of the house? | 1 | 2 | 3 | 4 |
| 4. | Do you need to stay in bed or a chair during the day? | 1 | 2 | 3 | 4 |
| 5. | Do you need help with eating, dressing, washing yourself or using the toilet? | 1 | 2 | 3 | 4 |
| Du | ring the past week: | Not at | A<br>Little | Quite<br>a Bit | Very<br>Much |
| 6. | Were you limited in doing either your work<br>or other daily activities? | 1 | 2 | 3 | 4 |
| 7. | Were you limited in pursuing your hobbies or other leisure time activities? | 1 | 2 | 3 | 4 |
| 8. | Were you short of breath? | 1 | 2 | 3 | 4 |
| 9. | Have you had pain? | 1 | 2 | 3 | 4 |
| 10. | Did you need to rest? | 1 | 2 | 3 | 4 |
| 11. | Have you had trouble sleeping? | 1 | 2 | 3 | 4 |
| 12. | Have you felt weak? | 1 | 2 | 3 | 4 |
| 13. | Have you lacked appetite? | 1 | 2 | 3 | 4 |
| 14. | Have you felt nauseated? | 1 | 2 | 3 | 4 |
| 15. | Have you vomited? | 1 | 2 | 3 | 4 |

Please go on to the next page


| Du | ring the past week: | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|---|
| 16. | Have you been constipated? | 1 | 2 | 3 | 4 |
| 17. | Have you had diarrhea? | 1 | 2 | 3 | 4 |
| 18. | Were you tired? | 1 | 2 | 3 | 4 |
| 19. | Did pain interfere with your daily activities? | 1 | 2 | 3 | 4 |
| 20. | Have you had difficulty in concentrating on things, like reading a newspaper or watching television? | 1 | 2 | 3 | 4 |
| 21. | Did you feel tense? | 1 | 2 | 3 | 4 |
| 22. | Did you worry? | 1 | 2 | 3 | 4 |
| 23. | Did you feel irritable? | 1 | 2 | 3 | 4 |
| 24. | Did you feel depressed? | 1 | 2 | 3 | 4 |
| 25. | Have you had difficulty remembering things? | 1 | 2 | 3 | 4 |
| 26. | Has your physical condition or medical treatment interfered with your <u>family</u> life? | 1 | 2 | 3 | 4 |
| 27. | Has your physical condition or medical treatment interfered with your <u>social</u> activities? | 1 | 2 | 3 | 4 |
| 28. | Has your physical condition or medical treatment caused you financial difficulties? | 1 | 2 | 3 | 4 |

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

# For the following questions please circle the number between 1 and 7 that best applies to you $\,$

 29. How would you rate your overall health during the past week?

 1
 2
 3
 4
 5
 6
 7

 Very poor
 Excellent

 30. How would you rate your overall quality of life during the past week?

 1
 2
 3
 4
 5
 6
 7

 Very poor
 Excellent


<sup>©</sup> Copyright 1995 EORTC Quality of Life Group. All rights reserved. Version 3.0

Table 1 EORTC QLQ-C30 Scoring Guide

| | Scal<br>e | Number of items | Item<br>range* | Version 3.0 Item numbers | Function scales |
|---|---|---|---|---|---|
| Global health status / QoL | | | | | |
| Global health status/QoL (revised)† | QL2 | 2 | 6 | 29, 30 | |
| <b>Functional scales</b> | | 1 | l | l | 1 |
| Physical functioning (revised)† | PF2 | 5 | 3 | 1 to 5 | F |
| Role functioning (revised)† | RF2 | 2 | 3 | 6, 7 | F |
| Emotional functioning | EF | 4 | 3 | 21 to 24 | F |
| Cognitive functioning | CF | 2 | 3 | 20, 25 | F |
| Social functioning | SF | 2 | 3 | 26, 27 | F |
| Symptom scales / items | | l | l . | I | I |
| Fatigue | FA | 3 | 3 | 10, 12, 18 | |
| Nausea and vomiting | NV | 2 | 3 | 14, 15 | |
| Pain | PA | 2 | 3 | 9, 19 | |
| Dyspnoea | DY | 1 | 3 | 8 | |
| Insomnia | SL | 1 | 3 | 11 | |
| Appetite loss | AP | 1 | 3 | 13 | |
| Constipation | СО | 1 | 3 | 16 | |
| Diarrhoea | DI | 1 | 3 | 17 | |
| Financial difficulties | FI | 1 | 3 | 28 | |

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

#### **Scoring Algorithm**

The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.

The principle for scoring these scales is the same in all cases:

1. Estimate the average of the items that contribute to the scale; this is the raw score.


<sup>\*</sup> *Item range* is the difference between the possible maximum and the minimum response to individual items; most items take values from 1 to 4, giving *range* = 3.

<sup>† (</sup>revised) scales are those that have been changed since version 1.0, and their short names are indicated in this manual by a suffix "2" – for example, PF2.

2. Use a linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

The technical details are provided below.

If items  $I_1, I_2, ... I_n$  are included in a scale, the procedure is as follows:

Calculate the raw score (RS) as follows: RS= $(I_1+I_2+...+I_n)/n$ 

Apply the linear transformation as follows:

- Functional scales: Scale score =  $(1 ((RS 1)/range) \times 100$
- Symptom scales / items: Scale score =  $(RS 1)/range \times 100$
- Global health status/QoL: Scale score =  $(RS 1)/range \times 100$

where Range is the difference between the maximum possible value of RS and the minimum possible value. The QLQ-C30 has been designed so that all items in any scale take the same range of values. Therefore, the range of RS equals the range of the item values (see Table 1).

If at least half the components of a scale are present, then the scale score will be calculated using the average of all items answered as the raw score; otherwise the score will be set to missing. For single measures, if the item is missing, the scale score is set to missing.


# 2. The Medical Outcomes Study-Short Form-36 (SF-36)

| ■<br> | Subject ID | Quality of Life CLL III Study SF-36 (page 1 of 3) riews about your health. This information will help you keep tra | | | | ssessment |
|---|---|---|---|---|---|---|
| an | d how well you are able to conduct y | our daily ac | tivities. | | | |
| | swer every questions by selecting t<br>estion, please give the best answer | | | | | wer a |
| 1. | In general, would you say your health | is: O Excelle | nt O Very | good O Good | I O Fair | O Poor |
| 2. | Compared to one year ago, how woul you rate your health, in general, now? | | - | what O About now the same | <ul><li>Somewhat worse now</li></ul> | • |
| Do | es your health limit you in the activi | ties listed be | low? If so, ho | w much? | | |
| | | Yes, limited<br>a lot | Yes, limited<br>a little | No, not<br>limited at all | | |
| 3. | Vigorous activities, such as running, lifting heavy objects, or participating in strenuous sports? | 0 | 0 | 0 | | |
| 4. | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf? | 0 | 0 | 0 | | |
| 5. | Lifting or carrying groceries? | 0 | 0 | 0 | | |
| 6. | Climbing several flights of stairs? | 0 | 0 | 0 | | |
| 7. | Climbing one flight of stairs? | 0 | 0 | 0 | | |
| 8. | Bending, kneeling, or stooping? | 0 | 0 | 0 | | |
| 9. | Walking more than a mile? | 0 | 0 | 0 | | |
| 10 | ). Walking several blocks? | 0 | 0 | 0 | | |
| 11 | . Walking one block? | 0 | 0 | 0 | | |
| 12 | 2. Bathing or dressing yourself? | 0 | 0 | 0 | | 46547 |

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021


| Subject ID Quality CLL III SF-36 (page | Study | | Assessment |
|---|---|---|---|
| During the PAST 4 WEEKS, have you had any of the following problems with your work or other regular activities as a result of your PHYSICAL HEALTH? | | | |
| 13. Cut down on the amount of time you spent on work or other activities? | O Yes | O No | |
| 14. Were limited in the kind of work or other activities? | O Yes | O No | |
| 15. Accomplished less than you would like? | O Yes | O No | |
| 16. Had difficulty performing the work or other activities (e.g., it took extra effort)? | O Yes | O No | |
| <ul><li>17. Cut down on the amount of time you spent on work or other activities?</li><li>18. Accomplished less than you would like?</li></ul> | O Yes | O No | |
| I did not do work or other activities as carefully as usual. | | ○ False | |
| 20. During the PAST 4 WEEKS, to what extent have your P normal social activities with family, friends, neighbors, or O Not at all O A little bit O Moderate | r groups? | HEALTH or EM | MOTIONS interfered with your |
| 21. How much bodily pain did you have during the PAST 4 | WEEKS? | | |
| O None O Very mild O Mild O Mo | derate | O Severe | O Very severe |
| 22. During the PAST 4 WEEKS, how much did pain interferent and housework)? | e with your | normal work ( | including work outside the ho |
| O Not at all O A little bit O Moderate | ly ( | Quite a bit | O Extremely |

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021


| CL | ality of L | dy | | | Assessi | ment |
|---|---|---|---|---|---|---|
| For each question, please indicate the one answer | r that come | | to the way | you have | been feelin | g in the |
| PAST 4 WEEKS | | | | and the second s | | |
| During the PAST 4 WEEKS, how much of the time. | | | | | | |
| | All of the time | Most of the time | A good bit of the time | Some of the time | A little bit of the time | None of the time |
| 23. Did you feel full of pep? | 0 | 0 | 0 | 0 | 0 | 0 |
| 24. Have you been a very nervous person? | 0 | 0 | 0 | 0 | 0 | 0 |
| 25. Have you felt so down in the dumps that nothing could cheer you up? | 0 | 0 | 0 | 0 | 0 | 0 |
| 26. Have you felt calm and peaceful? | 0 | 0 | 0 | 0 | 0 | 0 |
| 27. Did you have a lot of energy? | 0 | 0 | 0 | 0 | 0 | 0 |
| 28. Have you felt downhearted and blue? | 0 | 0 | 0 | 0 | 0 | 0 |
| 29. Did you feel worn out? | 0 | 0 | 0 | 0 | 0 | 0 |
| 30. Have you been a happy person? | 0 | 0 | 0 | 0 | 0 | 0 |
| 31. Did you feel tired? | 0 | 0 | 0 | 0 | 0 | 0 |
| 32. Has your HEALTH limited your social activities (like visiting friends or close relatives, etc.)? | 0 | 0 | 0 | 0 | 0 | 0 |
| Please choose how TRUE or FALSE these statement | ents are for | r you. | | | | |
| | Definitely true | Mostly true | Not<br>sure | Mostly false | Definitely false | |
| 33. I seem to get sick a little easier than other people. | . 0 | 0 | 0 | 0 | 0 | |
| 34. I am as healthy as anyone I know. | 0 | 0 | 0 | 0 | 0 | |
| 35. I expect my health to get worse. | 0 | 0 | 0 | 0 | 0 | |
| 36. My health is excellent. | 0 | 0 | 0 | 0 | 0 | |

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021


Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

| ITEMS | SCALES | Dime | nsions |
|---|---|---|---|
| 3. Vigorous activities | | | |
| 4. Moderate activities | | | |
| 5. Lift, carry groceries | | | |
| 6. Climb several flights | Scale 1: | | |
| 7. Climb one flight | Physical Functioning | | |
| 8. Bend, kneel | (PF) | | |
| 9. Walk mile | | | |
| 10. Walk several blocks | | | |
| 11. Walk one block | | | |
| 12. Bathe, dress | | Dimension A: PHYSICAL HELTH | |
| 13. Cut down time | | 3 5 | |
| 14. Accomplished less | Scale 2: | SIC | |
| 15. Limited in kind | Role-Physical (RP) | AL | |
| 16. Had difficulty | | HOH | |
| 21. Pain-magnitude | Scale 3: | EL A: | |
| 22. Pain-interfere | Bodily Pain (BP) | | |
| General health rating | | | |
| 36. Excellent | Scale 4: | | |
| 34. As healthy as anyone | General Health (GH) | | |
| 33. Sick easier | | | |
| 35. Health worse | | | |
| 23. Pep/life | | | |
| 27. Energy | Scale 5: | | [ ≦ |
| 29. Worn out | Vitality (VT) | İ | |
| 31. Tired | | | Dimension B:<br>MENTAL HEALTH |
| 32 Social-extent | Scale 6: | | L |
| 20. Social-time | Social Functioning (SF) | | |
| 17. Cut down time | | | ₽.Β. |
| 18. Accomplished less | Scale 7: | | 🗄 |
| 19. Not careful | Role-Emotional (RE) | | |
| 24. Nervous | | | |
| 25. Down in dumps | Scale 8: | | |
| 26. Peaceful | Mental Health (MH) | | |
| 28. Blue/sad | | | |
| 30. Нарру | | | |
| 2. Change in reported health | | ' | |


#### **Appendix F: Adverse Events of Clinical Interest**

Below please see the definition and searching criteria for adverse events of clinical interest.

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

# Definition of Adverse Event of Special Interest and Events of Clinical Interest (MedDRA version 24.0)

#### 1. Adverse Event of Special Interest (AESI)

The following preferred terms (PT) for the ventricular arrhythmias AESI include:

- Torsade de pointes
- Ventricular arrhythmia
- Ventricular extrasystoles
- Ventricular fibrillation
- Ventricular flutter
- Ventricular tachyarrhythmia
- Ventricular tachycardia

#### 2. Events of Clinical Interest

The Events of Clinical Interest (ECIs) have been identified based on preclinical findings, emerging data from clinical studies relating to acalabrutinib, and pharmacological effects of approved Bruton's tyrosine kinase (BTK) inhibitors. The adverse events (AEs) selected for dedicated analysis were evaluated using Standardized MedDRA Queries (SMQs), where available, by System Organ Classes (SOCs), or by Sponsor-defined baskets of MedDRA Adverse Event Grouped Terms.

| Category | Subcategory | Definition |
|----------------|---------------------|------------------------|
| Cardiac events | | SOC Cardiac disorders |
| | Atrial fibrillation | PT Atrial fibrillation |
| | | PT Atrial flutter |


| | Ventricular | PT Torsade de pointes |
|---|---|---|
| | tachyarrhythmias | <ul> <li>PT Ventricular fibrillation</li> </ul> |
| | | PT Ventricular flutter |
| | | PT Ventricular tachyarrhythmia |
| | | PT Ventricular tachycardia |
| Cytopenias – | | • SMQ Haematopoietic erythropenia [narrow + |
| Anemia | | broad] |
| Cytopenias – | | SMQ Haematopoietic leukopenia [narrow + |
| Leukopenia | | broad] |
| | Neutropenia | PT Band Neutrophil count decreased |
| | | PT Band neutrophil percentage decreased |
| | | PT Cyclic neutropenia |
| | | PT Febrile Neutropenia |
| | | PT Idiopathic neutropenia |
| | | PT Neutropenia |
| | | PT Neutropenic infection |
| | | PT Neutropenic sepsis |
| | | PT Neutrophil count decreased |
| | | PT Neutrophil percentage decreased |
| | Other leukopenia | SMQ Haematopoietic leukopenia [narrow + |
| | | broad] excluding PTs for neutropenia above |
| Cytopenias - | | SMQ Haematopoietic thrombocytopenia |
| Thrombocytopenia | | [narrow + broad] |
| Hemorrhage | | SMQ Haemorrhage terms (excl laboratory |
| | | terms) |
| | Major hemorrhage | • As per definition (see Section 3 below) |
| | Other leukopenia | <ul> <li>PT Neutrophil percentage decreased</li> <li>SMQ Haematopoietic leukopenia [narrow +</li> </ul> |
| | | broad] excluding PTs for neutropenia above |
| Cytopenias - | | SMQ Haematopoietic thrombocytopenia |
| Thrombocytopenia | | [narrow + broad] |
| Hemorrhage | | SMQ Haemorrhage terms (excl laboratory |
| | | terms) |
| | Major hemorrhage | • As per definition (see Section 3 below) |

Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021


| Hepatotoxicity | | • | SMQ [narrow] Hepatic failure, fibrosis and |
|---|---|---|---|
| | | | cirrhosis and other liver damage-related |
| | | | conditions |
| | | • | SMQ [narrow] Hepatitis, non-infectious |
| | | • | SMQ [narrow] Liver related investigations |
| | | | signs |
| Hypertension | | • | SMQ Hypertension [narrow] |
| Infections | | • | SOC Infections and infestations |
| Interstitial lung | | • | SMQ [narrow] Interstitial lung disease |
| disease/Pneumonitis | | | |
| Second primary | | • | SMQ Malignant tumours (including |
| malignancies | | | Haematological malignant tumours SMQ and |
| | | | Non-haemoatological malignant tumours |
| | | | SMQ) |
| | | • | SMQ Malignant lymphomas [narrow] |
| | | | SMQ Myelodysplastic syndrome [narrow] |
| | Second primary | • | The above excluding PTs mapping to HLT |
| | malignancies | | Skin neoplasms malignant and unspecified |
| | (excluding non | | (excluding melanoma) |
| | melanoma skin) | | |
| Tumor lysis | | • | PT Tumour lysis syndrome |
| syndrome | | | |

Protocol: ACE-CL-003

Amendment 1: 06 Oct 2021

AE=adverse event; ALT=alanine aminotransferase; AST=aspartate aminotransferase; HLT=high-level term; ISS=integrated safety summary; PT=preferred term; SAE=serious adverse event; SMQ=Standardised MedDRA Query; ULN=upper limit of normal. MedDRA version 24.0


Protocol: ACE-CL-003 Amendment 1: 06 Oct 2021

